CLINICAL TRIAL: NCT03375398
Title: Determination of the Postprandial Glucose And Insulin Responses of White Rice Alone And White Rice Consumed With Sugardown™
Brief Title: Determination of the PPG and Insulin Responses of Rice Alone and Rice Consumed With Sugardown™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: PAZ320-001
Record Dates: First submitted 2014-02-11; First posted 2017-12-18 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Postprandial Hyperglycemia
Keywords: SUGARDOWN™; Galactomannan; Postprandial blood glucose; Insulin
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance | interventions — PAZ320

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 3 tablets Sugardown™ (Experimental): Repeated-measures, open cross-over design: 10 subjects consumed three different test meals comprising of white rice consumed with 3 tablets Sugardown™
  Interventions: Dietary Supplement: Sugardown™
- Rice only (Placebo Comparator): Repeated-measures, open cross-over design: 10 subjects consumed three different test meals comprising of white rice
  Interventions: Dietary Supplement: Rice
- 6 tablets Sugardown™ (Experimental): Repeated-measures, open cross-over design: 10 subjects consumed three different test meals comprising of white rice consumed with 6 tablets Sugardown™
  Interventions: Dietary Supplement: Sugardown™

INTERVENTIONS:
Dietary Supplement: Rice — Test food #1: White Rice <63.0 g (dry) Jasmine rice consumed together with 250 mL water
  Other Names: BTI320; PAZ320
  Arms: Rice only
Dietary Supplement: Sugardown™ — Test food #2: White Rice < 63.0 g (dry) Jasmine rice + 3 Sugardown™ tablets consumed together with 250 mL water Test food #3: White Rice < 63.0 g (dry) Jasmine rice + 6 Sugardown™ tablets consumed together with 250 mL water
  Other Names: BTI320; PAZ320
  Arms: 3 tablets Sugardown™; 6 tablets Sugardown™

SUMMARY:
This study was a partly controlled laboratory-based study comparing the short-term postprandial blood glucose and insulin responses produced by 3 test meals containing white rice alone or with SUGARDOWN™ (Galactomannan) in overweight adults.

DETAILED DESCRIPTION:
STUDY SUMMARY This study was a partly controlled laboratory-based study comparing the short-term postprandial blood glucose and insulin responses produced by three test meals containing white rice alone or with SUGARDOWN™ (Galactomannan) in overweight adults. In the study, subjects were their own controls. Effects of the two test meals containing SUGARDOWN™ were compared to the effects produced by test meals containing an equal-carbohydrate portion of white rice alone (the control meal). The study used a repeated-measures design, such that every subject consumed each meal on two separate occasions, completing a total of six separate test sessions. Each subject completed their test sessions on separate weekday mornings at a similar time of day, as close as possible to the time they would normally eat breakfast.

SUBJECTS Ten healthy, non-smoking, overweight or obese subjects (4 females, 6 males) voluntarily participated in this study. The mean ± SD age of the subjects was 29.2 ± 3.3 yr (range: 25.6 - 36.8 yr), and their mean ± SD body mass index value was 27.3 ± 1.1 kg/m2 (range: 25.5 - 28.7 kg/m2).

Volunteers were given detailed written and verbal information about all of the study's inclusion criteria and experimental procedures. If the volunteers decided that they would like to participate in the study, they were asked to come to the research centre on another morning, where they completed a detailed screening questionnaire that assessed their current health status and medical history. In order to participate in the study, the volunteers had to meet the inclusion criteria listed below. All suitable volunteers that were invited to participate in the study were required to sign a detailed subject information sheet and a consent form before commencing any experimental procedures.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 25-65 years.
* Non-smoker.
* Stable body weight within the overweight weight range for their height (BMI values > 25 kg/m2).
* Normal dietary habits; not dieting or eating in an overly restrictive fashion in the past 3 months.
* A regular pattern of low to moderate physical activity.
* Able to fast for ≥ 10 hours the night before each test session.
* Able to refrain from eating a legume-based evening meal or drinking alcohol the day before each test session.
* Finds the test foods suitable for consumption within 12 minutes.
* Participant covered by social security or a similar system.
* Not taking any treatment for anorexia, weight loss, or any form of treatment or medication likely to interfere with metabolism or dietary habits.
* Signed the informed consent form for the study.

Exclusion Criteria:

* Currently following a restrictive diet (low-calorie, low-carbohydrate, vegan).
* Any clinically significant physical or mental illness.
* Suffering from a food allergy or serious food intolerance.
* Regularly taking prescription medication other than standard contraceptive medication.
* Females who are currently pregnant, breast-feeding, trying to become pregnant or not using an acceptable contraceptive.
* Participating in another clinical trial or participated in another clinical trial within the last week.
* Undergoing general anaesthesia in the month prior to inclusion.
* Subject in a situation, which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Postprandial increment glucose under the area curve (iAUC) | 2 days
  Blood samples were collected into a micro-centrifuge tube containing the anticoagulant, heparin sodium salt. Plasma glucose concentrations were measured in duplicate using a spectrophotometric centrifugal analyser employing the glucose hexokinase/glucose-6-phosphate dehydrogenase enzymatic assay.

SECONDARY OUTCOMES:
Postprandial increment insulin under the area curve (iAUC) | 2 days
  Each blood sample was collected into a micro-centrifuge tube containing the anticoagulant. Plasma insulin concentrations were measured using a solid phase antibody-coated tube radioimmunoassay kit.

CONTACTS AND LOCATIONS:
Overall Officials: Jennie Brand-Miller, Prof., Principal Investigator — Human Nutrition Unit School of Molecular Bioscience, University of Sydney, Australia